CLINICAL TRIAL: NCT01488734
Title: Bioavailability and Biological Effects of Vitamin D2 Contained in Mushroom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GCO 11-0899; 11-01366
Record Dates: First submitted 2011-12-06; First posted 2011-12-08 (Estimated); Last update posted 2017-04-14 (Actual); Status verified 2017-04

CONDITIONS: Vitamin D Deficiency; Metabolic Syndrome; Prediabetes
Keywords: Vitamin D; Mushroom; Cholecalciferol; Prediabetes; Metabolic Syndrome
MeSH Terms: conditions — Vitamin D Deficiency; Metabolic Syndrome; Prediabetic State | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mushroom with 600 IU vitamin D2 (Experimental): Mushroom with 600 IU of vitamin D2 daily and placebo tablet
  Interventions: Dietary Supplement: Mushroom with 600 IU vitamin D2; Drug: Placebo
- Mushroom with 4000 IU Vitamin D2 (Experimental): Mushroom with 4000 IU of Vitamin D2 daily and placebo tablet
  Interventions: Dietary Supplement: Mushroom with 4000 IU Vitamin D2; Drug: Placebo
- 600 IU Vitamin D3 and untreated mushroom (Active Comparator): Commercially available tablets with 600 IU/day of Vitamin D3 and untreated mushroom
  Interventions: Dietary Supplement: 600 IU Vitamin D3 and untreated mushroom
- 4000 IU Vitamin D3 and untreated mushroom (Active Comparator): Commercially available tablets with 4000 IU/day of Vitamin D3 and untreated mushroom
  Interventions: Dietary Supplement: 4000 IU Vitamin D3 and untreated mushroom

INTERVENTIONS:
Dietary Supplement: Mushroom with 600 IU vitamin D2 — Subjects in this group will eat daily meals containing mushrooms fortified with 600 IU of Vitamin D2. These subjects will also take one placebo tablet per day.
  Arms: Mushroom with 600 IU vitamin D2
Dietary Supplement: Mushroom with 4000 IU Vitamin D2 — Subjects in this group will eat daily meals containing mushrooms fortified with 4000 IU of Vitamin D2. These subjects will also take one placebo tablet per day.
  Arms: Mushroom with 4000 IU Vitamin D2
Dietary Supplement: 600 IU Vitamin D3 and untreated mushroom — Subjects in this group will take one commercially available tablet of 600 IU of Vitamin D3. These subjects will also eat one meal per day with untreated (inactive) mushrooms.
  Arms: 600 IU Vitamin D3 and untreated mushroom
Dietary Supplement: 4000 IU Vitamin D3 and untreated mushroom — Subjects in this group will take one commercially available tablet of 4000 IU of Vitamin D3. These subjects will also eat one meal per day with untreated (inactive) mushrooms.
  Arms: 4000 IU Vitamin D3 and untreated mushroom
Drug: Placebo — Placebo for the fortified mushroom arms
  Arms: Mushroom with 4000 IU Vitamin D2; Mushroom with 600 IU vitamin D2

SUMMARY:
The purpose of this study is to compare the safety and efficacy of two different amounts of vitamin D2 (600 or 4000 International Units/day) provided by mushrooms added to one of the daily meals versus same doses of vitamin D3 provided as oral supplements sold in any drugstore in reaching adequate or optimal blood levels of 25(OH)D in people with Vitamin D deficiency and pre-diabetes (high blood sugar without full blown diabetes) or the metabolic syndrome. Metabolic syndrome is the name of a group of risk factors that raise the risk for heart disease and other health problems, such as diabetes and stroke as described by the US department of Health and Human Services.

This study will also attempt to demonstrate and compare the effect of the intervention with above two doses of vitamin D on blood levels of tests that show inflammation.

DETAILED DESCRIPTION:
Poor vitamin D status is now considered epidemic in North America. In addition to its effects on bone metabolism, Vitamin D has several other important biological effects including modulating the immune system, stimulating the production of insulin and decreasing renin production in the kidney. Furthermore, the active metabolite of vitamin D, 1,25 dihydroxyvitamin D (1,25(OH)2D), is a very potent inhibitor of cellular proliferation and inducer of terminal differentiation and vitamin D deficiency has been associated with higher prevalence of cancer, autoimmune diseases, including multiple sclerosis, rheumatoid arthritis, type 1 diabetes and hypertension.

The current recommendations for dietary vitamin D in North America are much too low to maintain optimal levels of 25(OH)D associated with disease prevention. The majority of circulating 25(0H) D originates from cutaneous synthesis upon exposure to adequate sunlight. However, seasonal changes, living at high latitudes or low polluted altitudes, dark skin pigmentation and aging are among the many factors that can impede this process requiring periodic reliance on dietary sources to supply the precursor to 25(OH)D.

In November of 2010, the Institute of Medicine (IOM) of the National Academy of Science established new DRI values for vitamin: EAR (Estimated Average Requirement) of 400 IU (10 µg; RDA ( Recommended Daily Intake) of 600 IU (15µg) for adults up to 70 years of age, and an UL of 4000 IU (50µg) (21). The IOM also discourages the taking of dietary supplements to achieve the RDA for vitamin D and encourages Americans to achieve their needed vitamin D through food sources.

The proposed study will be to provide meals with one serving of fresh mushroom per day that could have two different levels of vitamin D2 in it (600 IU or 4,000 IU/day, which are the 2011 currently recommended RDA to age 70 AI and UL, respectively) for four months and test both the bioavailability of vitamin D in mushroom, as reflected in blood 25(OH)D levels, as well as the effect of vitamin D on markers of disease (e.g. C-reactive protein (CRP), Hemoglobin A1c, etc). The vitamin D2 amount in mushrooms can easily be manipulated just by adjusting the time and distance of their UVB exposure. Two groups will be compared with controls who will receive the same dose of vitamin D3 in the form of tablets commercially available (600 IU or 4000 IU/day).

ELIGIBILITY:
Inclusion Criteria:

* Adult non-smoking subjects from ages 30 to 90, any race or gender
* Presence of at least two of the following characteristics:

  * Waist circumference:

Men: > 102 cm Women: > 88 cm

* Blood pressure: > 130/85 mm Hg (or use of anti-BP medication)
* HDL-cholesterol:

Men: < 40 mg/dL Women: < 50 mg/dL

* Triglycerides: > 150 mg/dL (or use of medications for high triglycerides such as fibrates or nicotinic acid)
* Fasting blood sugar > 100 mg/dl (or use of metformin), but a HbA1c < 6.5%

Exclusion Criteria:

* Blood levels of 25(OH)D > 50 nmol/L
* Regular intake of vitamin D fortified milk exceeding approximately 3 glasses/day
* Lack of the ability to comprehend instructions and/or sign the consent form
* Inability to comply with the potential requirement to eat a daily portion of provided mushroom together with meals
* Inability to comply with the rule of avoiding any beach days during the duration of the study
* Any projected trip to sunny places such as Puerto Rico and the Caribbean during the period of study
* Any attendance to tanning studios during the period of study
* Women who regularly use a veil over their heads
* Any history of kidney stone formation
* Non-traumatic bone fracture over the past 3 years
* Any form of vitamin D supplement intake, including combined calcium and vitamin D products
* Active smoking

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
25OH Vitamin D level | at 4 months
  To compare the efficacy of two different doses of vitamin D2 (600 or 4000 IU/day) provided by Vitamin D2 fortified mushrooms added to one of the daily meals versus same doses of vitamin D3 provided as oral supplements in reaching adequate or optimal circulating levels of 25(OH) D in a racially diverse group of subjects with Vitamin D deficiency and pre-diabetes or the metabolic syndrome.

SECONDARY OUTCOMES:
Serum calcium | at 1 month
  To assess the safety of the intervention with respect to serum calcium levels in all study subjects. Measured at each study visit (1, 2, 3, and 4 months)
Serum calcium | at 2 months
  To assess the safety of the intervention with respect to serum calcium levels in all study subjects. Measured at each study visit (1, 2, 3, and 4 months)
Serum calcium | at 3 months
  To assess the safety of the intervention with respect to serum calcium levels in all study subjects. Measured at each study visit (1, 2, 3, and 4 months)
Serum calcium | at 4 months
  To assess the safety of the intervention with respect to serum calcium levels in all study subjects. Measured at each study visit (1, 2, 3, and 4 months)
Markers of inflammation and metabolic control | at 4 months
  To demonstrate and compare the effect of the intervention with above two doses of vitamin D on circulating levels of markers of inflammation and metabolic control (CRP, tumor necrosis factor (TNF), hemoglobin A1c, insulin, blood glucose, lipids).

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Uribarri, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States